CLINICAL TRIAL: NCT06353646
Title: Efficacy and Safety Trial of XH001 (Neoantigen Cancer Vaccine) Sequential Combination With Immunocheckpoint Inhibitor and Chemotherapy in Adjuvant Therapy for Patients With Resected Pancreatic Cancer
Brief Title: XH001 Combination With Immunocheckpoint Inhibitor and Chemotherapy for Patients With Resected Pancreatic Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wu Wenming (Other)
Collaborators: NeoCura (Industry)
Responsible Party: Sponsor-Investigator, Wu Wenming, Prof., Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XKY-C-004
Record Dates: First submitted 2024-03-28; First posted 2024-04-09 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Pancreatic Cancer
Keywords: cancer vaccine, mRNA, neoantigen; Pancreatic Cancer; adjuvant therapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Ipilimumab; sintilimab; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Experimental): XH001;Ipilimumab Injection;Chemotherapy
  Interventions: Biological: XH001; Drug: Ipilimumab Injection; Drug: Chemotherapy
- Arm B (Experimental): XH001;Sintilimab Injection;Chemotherapy
  Interventions: Biological: XH001; Drug: Sintilimab injection; Drug: Chemotherapy

INTERVENTIONS:
Biological: XH001 — XH001 will be administered 12 weeks post-tumor resection (+/- 2 weeks)
Drug: Ipilimumab Injection — Ipilimumab will be administered 12 weeks post-tumor resection (+/- 2 weeks)
  Arms: Arm A
Drug: Sintilimab injection — Sintilimab will be administered 12 weeks post-tumor resection (+/- 2 weeks)
  Arms: Arm B
Drug: Chemotherapy — gemcitabine + capecitabine

SUMMARY:
This is a single-center, open label, single-arm, investigator-initiated study to evaluate the efficacy and safety of XH001 (neoantigen cancer vaccine) sequential combination with immunocheckpoint inhibitor and chemotherapy in pancreatic cancer patients following surgical resection.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form;
* Aged 18 to 75 years old;
* Histologically or cytologically confirmed diagnosis of pancreatic adenocarcinoma;
* Completed an R0 or R1 surgical resection as determined by pathology；
* Have not received any prior neoadjuvant therapy;
* ECOG score is 0 or 1;
* Life expectancy of greater than 12 months;
* CA19-9 <100U/mL before initial chemotherapy;
* Patients must have adequate organ and marrow function defined by study-specified laboratory tests prior to initial study drug.
* Woman of childbearing potential must have a negative pregnancy test and follow contraceptive guidelines as defined per protocol.

Exclusion Criteria:

* Borderline resectable pancreatic cancer;
* Evidence of disease recurrence or metastasis following surgical resection at any time;
* Evidence of malignant ascites;
* Pre-existing inflammatory bowel disease or the presence of complete or partial bowel obstruction, or persistent severe diarrhea after surgery;
* Needs to receive long-term systemic anti-allergic drug or known hypersensitivity to any component of the study treatment;
* History of autoimmune disease;
* New cerebrovascular accident (including ischemic stroke, hemorrhagic stroke, and transient ischemic attack) within 6 months before screening;
* Acute myocardial infarction within 6 months before screening, or uncontrolled angina, uncontrolled arrhythmia, severe heart failure (see Appendix 3, New York Heart Association Heart Failure Classification Criteria NYHA Class ≥ III) and other cardiovascular diseases;
* Received immunomodulatory medications within 4 weeks prior to the date of the first dose (D1) of XH001, including but not limited to: IL-2, CTLA-4 inhibitors, CD40 agonists, CD137 agonists, IFN-α;
* Received blood transfusion, erythropoietin (EPO), granulocyte colony-stimulating factor (G-CSF) or granulocyte-macrophage colony-stimulating factor (GM-CSF) within 7 days prior to the first dose of XH001;
* Received therapeutic tumor vaccines;
* With congenital or acquired immunodeficiency;
* Participating in other clinical trials and not enrolled at the screening period;
* Unable or unwilling to comply with the study protocol due to potential health, mental or social conditions in the opinion of the investigator;
* Other conditions that, in the opinion of the investigator, would make participation in this study inappropriate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
DFS | up to 36 months
  disease-free survival (DFS)
DFS rate | up to 36 months
  disease-free survival rate
MFS | up to 36 months
  metastasis-free survival (MFS)
OS | From date of recruitment until the date of first documented date of death from any cause, assessed up to 36 months
  overall survival (OS)

SECONDARY OUTCOMES:
Elispot | up to 36 months
  Antigen-specific T-cell responses in peripheral blood
Adverse Event | up to 36 months
  Incidence and severity of adverse events (AEs), clinically significant abnormal changes in laboratory tests or other examinations (based on the Criteria for the Evaluation of Adverse Events [CTCAE] v5.0).
ctDNA | up to 36 months
  Changes of ctDNA compared to baseline
CA19-9 | up to 36 months
  Changes of CA19-9 compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Wenming WU, Prof., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No